CLINICAL TRIAL: NCT00354666
Title: A Randomised, Double-blind, Placebo-controlled, Dose Ascending Crossover Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Inhaled GSK159797 Delivered by Dry Powder Inhaler in Mild to Moderate Asthmatic Subjects
Brief Title: Single Doses GSK159797 On Patient Safety And Lung Function In Patients With Mild To Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2E101312
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: inhaled; asthmatic subjects; GSK159797; safety and tolerability; efficacy; dry powder
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

INTERVENTIONS:
Drug: GSK159797

SUMMARY:
This study was designed to test safety aspects and effects on lung function of a new dry powder version of GSK159797 for asthmatic subjects to inhale. This will allow comparison with previous studies which have only used inhalation of the drug as a vapour.

ELIGIBILITY:
Inclusion criteria:

* Subjects with mild to moderate stable asthma but no other lung problems.
* Male subjects or females who are not able to get pregnant (e.g. post-menopausal or surgically sterile).
* Non-smokers.
* Subjects that show a measurable improvement in the function of their lungs after a single dose of salbutamol.

Exclusion criteria:

* Any significant illness.
* Subjects with heart problems.
* Subjects who have had a cold or chest infection 2-4 weeks prior to the study.
* Subjects who take medication for their asthma, or other conditions, not compatible with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-09; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability including blood test results, effects on the heart, pulse rate and blood pressure, and side effects.

SECONDARY OUTCOMES:
Effects on the lung at 12 and 24hrs Effects on the heart, blood pressure and pulse rate at 8hrs Changes in the amount of glucose and potassium in the blood 4 and 8hrs Amount of drug in the body (blood and urine).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: B2E101312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2E101312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2E101312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2E101312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2E101312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register